CLINICAL TRIAL: NCT03333538
Title: A Double-blind Randomized Placebo-controlled Study of Safety and Immunogenicity of Medicinal Product GamEvac-Lyo, Vector-Based Vaccine Against Ebola Virus Disease, Lyophilisate for Preparation of Solution for Intramuscular Injection
Brief Title: A Double-blind Randomized Placebo-controlled Study of Safety and Immunogenicity of GamEvac-Lyo
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Research Institute of Influenza, Sankt-Peterburg, Russian Federation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01-GamEvac-Lyo-2017
Record Dates: First submitted 2017-09-29; First posted 2017-11-07 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
Keywords: Hemorrhagic Fever, Ebola; Ebola Virus Disease; Ebola Virus Vaccines; Hemorrhagic Fevers, Viral; GP protein, Ebola virus; Filoviridae Infections; RNA Virus Infections
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral; Filoviridae Infections; RNA Virus Infections

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: This clinical trial is designed as a double blind randomized placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1 (component A) (Experimental): a single administration of component A (VSV) of vaccine
  Interventions: Biological: GamEvac-Lyo (component A)
- Stage 1 (component B) (Experimental): a single administration of component B (Ad5) of vaccine
  Interventions: Biological: GamEvac-Lyo (component B)
- Stage 2 (Primary Group) (Experimental): 150 people who will receive the vaccine in the therapeutic scheme: the sequential introduction of components A and B with an interval of 21 days
  Interventions: Biological: GamEvac-Lyo
- Stage 2 (Controll Group) (Placebo Comparator): 50 people who will receive placebo in the therapeutic scheme: the sequential introduction of components A (placebo) and B (placebo) with an interval of 21 days
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GamEvac-Lyo (component A) — Biological: GamEvac-Lyo (vaccine) vaccination, single administration, component A
  Arms: Stage 1 (component A)
Other: Placebo — Placebo vaccination
  Arms: Stage 2 (Controll Group)
Biological: GamEvac-Lyo (component B) — Biological: GamEvac-Lyo (vaccine) vaccination, single administration, component B
  Arms: Stage 1 (component B)
Biological: GamEvac-Lyo — Biological: GamEvac-Lyo (vaccine) vaccination, therapeutic scheme: the sequential introduction of components A and b with an interval of 21 days
  Arms: Stage 2 (Primary Group)

SUMMARY:
The purpose of this study is to evaluate immunogenicity and safety of medicinal product GamEvac-Lyo- Vector-Based Vaccine against Ebola Virus Disease

DETAILED DESCRIPTION:
This clinical trial is designed as a double blind randomized placebo-controlled study to evaluate immunogenicity of medicinal product GamEvac-Lyo- Vector-Based Vaccine against Ebola Virus Disease The study will consist of two stages. At the first stage in this research is planned to study the safety and tolerability of one dose of component A and B combined vaccine vector against Ebola in 20 healthy volunteers: 10 for component A and 10 to component B. In the first stage, the placebo will not be used. The duration of screening up to 10 days.

Volunteers at the first stage will receive the drug 1 time on the first day of the study. On the third day of the study (48 hours after administration of the vaccine) they will be discharged from the hospital. There will also be 1 outpatient visit on day 7 after drug administration.

After interim analysis of safety data is subject to the consent of the local ethics Committee of the Research Centre about the possibility of further studies of the drug - will be started the second phase of the study, which, along with continued security research, provides the definition of the parameters of immunogenicity of the study drug. The second phase of the study will included 200 participants, including 150 people will receive the study drug and 50 will be a control group of observation - that is, will get a placebo.

Study Schedule Visit 0 (outpatient): screening Visit 1 (inpatient): Immunization with component A/placebo (observation at the hospital for 48 hours). Local adverse reactions will be monitored during the entire observation period; on the day of immunization - local and systemic reactions should be recorded 20 minutes, 5 and 8 hours after the vaccine administration. Later, in-hospital local and systemic adverse reactions to the product will be documented during physical examinations twice a day (morning and evening) and also prior the subjects are discharged from the hospital. Adverse events will be then recorded in the "Daily Diaries" kept by the subjects during the outpatient stage.

Visit 2: Day 7 after the first vaccine administration - outpatient setting. Visit 3 (inpatient) (Day 21) Immunization with component B/placebo (observation at the hospital for 48 hours): Local adverse reactions will be monitored during the entire observation period; on the day of immunization - local and systemic reactions should be recorded 20 minutes, 5 and 8 hours after the vaccine administration. Later, in-hospital local and systemic adverse reactions to will be documented during physical examinations twice a day (morning and evening) and also before the subjects are discharged from the hospital. Adverse events will be recorded in the "Daily Diaries" kept by the subjects during the outpatient stage.

Visits #4, 5, 6 - will be held in outpatient settings on Days 28 , 42 and 90 after the vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

* males and females within the age range from 18 to 55 years;
* written informed consent;
* subject body mass index (BMI): 18.5 ≤ BMI ≤ 30
* subject agrees to use effective contraceptive methods during the entire period of participation in the study (one of the following methods will be used: sexual abstinence; condoms (male or female with or without spermicidal agent); diaphragm or cervical cap with spermicidal agent; intrauterine device);
* absence of severe allergic diseases in the medical history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum disease)
* absence of allergic diseases relapses
* absence of acute infectious diseases/relapses of chronic diseases at the time of vaccine administration and 7 days prior to the vaccination
* no serious post-vaccination complications in patient's history following the earlier administration of immunobiological products
* in medical history and based on the screening results, subject has no diseases of the gastrointestinal system, liver, kidneys, cardiovascular system, CNS, locomotion system, urogenital and endocrine systems that could affect the assessment of the study results
* subject has a negative result of the blood or urine pregnancy test (for females of childbearing age)
* subject has negative tests for HIV, hepatitis B and С, syphilis
* subject has a negative result of the urine test for residual narcotic drugs
* subject has no hematopoietic malignancies
* subject has no malignant neoplasms
* indicators of complete blood count test at a screening visit are not heigher/lower from 1,1*ULN/LLN (upper limit of normal/lower limit of normal)
* indicators of clinical biochemical analysis at a screening visit: blood urea nitrogen, creatinine, glutamic-pyruvic transaminase, glutamate-oxaloacetate-transaminase, blood glucose test, creatinkinase, total protein, bilirubin are not heigher/lower from 1,1*ULN/LLN (upper limit of normal/lower limit of normal). Total cholesterol level from 3,6 mmol/L to 7,8 mmol/L.
* absence of inflammatory or dystrophic myocardial changes based on ECG data.
* absence of previous immunization with any vaccine against Ebola virus disease based on medical history data and during clinical trials as well

Exclusion Criteria:

* volunteer involvement in another study over the last 90 days

  * any immunization with vaccine over the last 30 days
  * presence of a concomitant illness in decompensation stage which might affect the course of the study (CNS organic lesion, decompensated cardiovascular diseases, any manifestations of kidney or acute liver failure, oncological diseases, diabetes mellitus)
  * subject has systolic blood pressure less than 100 mm Hg or greater than 139 mm Hg; diastolic blood pressure less than 60 mm Hg or greater than 90 mm Hg; heart rate lower than 60 beats per minute or above 90 beats per minute
  * any clinically significant laboratory abnormalities
  * subject has received treatment with steroids for the last 10 days
  * subject has received immunoglobulins or other blood products over the last 3 months
  * patient unwillingness to participate in the study
  * blood donation (at least 450 ml of blood or plasma) by subject in less than 2 months prior to the start of the study
  * subject has a history of the consumption of more than 5 units (0.25 l of pure alcohol) a week or drug abuse
  * subject smokes more than 10 cigarettes a day
  * positive results of urine test for narcotic drug residues
  * positive result of breath alcohol test (in the expired air sample)
  * subject has no ability to understand or follow the Protocol instructions
  * patient unwillingness to follow the procedures
  * pregnancy or breast feeding
  * subject has received immunosuppressive and/or immunomodulating agents within 6 months prior to the start of the study
  * history of regular injection or intranasal drug use; injection or intranasal drug use at the present time
  * subject has experienced symptoms of respiratory disease for the last 3 days
  * subject has exacerbation of allergic diseases or history of anaphylactic reactions or angioneurotic edema
  * previous history of hypersensitivity or allergic reactions to the administration of any vaccines
  * allergic reactions to the vaccine components

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants With Adverse Events
Number of Participants With Serious Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants With Serious Adverse Events
Number of Participants with Solicited Local and Systemic Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants with Solicited Local and Systemic Adverse Events
Antibody levels against the EBOV glycoprotein GP measured by an enzyme-linked immunosorbent assay (ELISA) | at days 0, 21, 42, 28 and 90
  Determination of antibody levels against the EBOV glycoprotein GP measured by an ELISA vs. baseline values and placebo

SECONDARY OUTCOMES:
Assessment of antigen-specific cell-mediated immune response | at days 0 and 28
  determination of specific T-cell- mediated response to Ebola virus proteins vs. baseline values and placebo
Neutralizing antibody levels measured by a virus-neutralization assay | at days 0 and 28
  Determination of the neutralizing antibody titer for a virus in virus neutralization reaction vs. baseline values and placebo
Change of the vital signs (systolic and diastolic blood pressure, heart rate, body temperature) after administration of the product | through the whole study, an average of 90 days
  Evaluation of the product safety by assessing its impact on the vital signs (systolic and diastolic blood pressure, heart rate, body temperature) in healthy volunteers after administration of the product in comparison to placebo
Change of the clinical laboratory test results after administration of the product | through the whole study, an average of 90 days
  Evaluation of the product safety by assessing its impact on the clinical laboratory test results in healthy volunteers after administration of the product in comparison with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Zubkova, MD, PhD, Principal Investigator — Research Institute of Influenza
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No